CLINICAL TRIAL: NCT03816644
Title: 5-Cog Battery to Improve Detection of Cognitive Impairment and Dementia
Brief Title: 5-Cog Battery for Detecting Cognitive Impairment and Dementia
Acronym: 5-Cog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2018-9140; UG3NS105565 (NIH)
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Dementia; Cognitive Impairment; Mild Cognitive Impairment; Neurocognitive Disorders
Keywords: Cognitive screening; Primary care; Dementia; Cognitive Impairment; Mild Cognitive Impairment
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Neurocognitive Disorders | interventions — Health Literacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-Cog (Experimental): The 5-Cog coupled with a decision tree is a simple, 5-minute procedure that will identify older persons with cognitive impairment in primary care settings, and flag them for further evaluation. The 5-Cog includes the Picture Memory Impairment Screen (PMIS), Motoric Cognitive Risk syndrome (MCR), and the Symbol Match test. The 5-Cog will be given after randomization and before the patients sees the physician. The 5-Cog will sort patients with 'cognitive impairment' from those with 'no cognitive impairment'. After completing the 5-Cog, the non-physician tester will send a message through the Electronic medical record (EMR) system to provide the physician with the 5-Cog results and guide the them through the follow-up based on the results.
  Interventions: Other: 5-Cog
- Health Literacy & Grip Assessment (Active Comparator): The 5 minute assessment includes the Short Assessment of Health Literacy (SAHL) and a grip assessment measured using a handgrip dynamometer. After completing the SAHL and grip assessment, the non-physician tester will send a message through the EMR to provide the physician with the results from the assessments and guide the them through the follow-up based on the results.
  Interventions: Other: Health Literacy & Grip Assessment

INTERVENTIONS:
Other: 5-Cog — The 5-Cog is a 5 minute cognitive screen which will identify patients with 'cognitive impairment' from those with 'no cognitive impairment'.
  Arms: 5-Cog
Other: Health Literacy & Grip Assessment — The health literacy and grip assessment will take approximately 5 minutes, and will test the patient's comprehension and pronunciation of health-related terms as well as strength in their dominant hand. The screen will sort out patients with 'low health literacy' and 'frail (low grip strength)' from those with normal health literacy and normal grip strength.
  Arms: Health Literacy & Grip Assessment

SUMMARY:
Despite the availability of numerous cognitive assessment tools, cognitive impairment related to dementia is frequently under-diagnosed in primary care settings. The investigators have developed a 5-minute cognitive screen (5-Cog) coupled with a decision tree to overcome the technical, cultural and logistic barriers of current cognitive screens to improve dementia care in primary care patients with cognitive concerns.

DETAILED DESCRIPTION:
Despite the availability of numerous cognitive assessment tools, cognitive impairment related to dementia is frequently under-diagnosed in primary care settings, and is a more prevalent problem among older African-Americans and Hispanics than among older whites. Missed detection delays treatment of reversible conditions as well as provision of support services and critical planning. To overcome the technical, cultural and logistic barriers of current cognitive screens and dementia care in primary care settings the investigators have developed a 5-minute cognitive screen (5-Cog) coupled with a decision tree to identify persons at high risk of developing dementia in multi-ethnic primary care populations.

The 5-Cog includes the Picture based Memory Impairment Screen (PMIS), Motoric Cognitive Risk syndrome (MCR), and a brief non-memory picture based test (Symbol Match). The cognitive assessment will sort patients with 'cognitive impairment' from those with 'no cognitive impairment'. It is coupled with a decision tree to guide clinicians through the follow up based on results of the 5-Cog.

The primary objective is to test the ability of the 5-Cog and decision tree paradigm to improve dementia care in primary care patients with cognitive concerns.

The investigators propose a single-blind, randomized clinical trial (RCT) in 1,200 older primary care patients with cognitive concerns who will be randomized to receive the 5-Cog (intervention group) or a 5-minute health literacy and grip assessment (active control group). Non-physicians will administer the intervention and control assessments in primary care sites and will provide results for both arms to the treating physician with a decision tree follow up guide based on the results of the assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 and older.
2. Presence of cognitive or memory concerns expressed by patient, caregiver, health care provider or other source who knows the patient.
3. Registered as patient at Montefiore Medical Center and have a primary care doctor appointment that day.
4. Able to hear and see well enough to complete intervention or control assessments.
5. English or Spanish speaking.

Exclusion Criteria:

1. Prior diagnosis of dementia or MCI as ascertained by ICD-10 codes or the documentation of prescription for anti-dementia medications in EMR. Patients with a diagnosis containing any of the following terms will be excluded:

   1. "Dementia"
   2. "Mild Cognitive Impairment"
   3. "Alzheimer's Disease"
   4. "Creutzfeldt-Jakob Disease"
   5. "Major Neurocognitive Disorder"
   6. "Minor Neurocognitive Disorder"

   Patients with any of the following medications documented in their EMR will be excluded (generic = brand):
   1. Donepezil = Aricept
   2. Memantine = Namenda
   3. Rivastigmine = Exelon
   4. Galantamine = Razadyne
   5. Donepezil and Memantine = Namzaric
2. Adults who are permanent residents of a nursing facility.
3. Patients who do not speak English or Spanish.
4. Patients who are not seeing a primary care physician at the clinic that day.
5. Patients who are blind or deaf or cannot hear loud voice even with hearing aids.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1201 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Verghese, MBBS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within 1 year of study completion.
Access Criteria: Data access requests will be reviewed by the PI and Steering Committee. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Malik R, Weiss EF, Gottesman R, Zwerling J, Verghese J. Picture-Based Memory Impairment Screen: Effective Cognitive Screen in Ethnically Diverse Populations. J Am Geriatr Soc. 2018 Aug;66(8):1598-1602. doi: 10.1111/jgs.15422. Epub 2018 May 29. PMID 29808583
- [Derived] Verghese J, Chalmer R, Stimmel M, Weiss E, Zwerling J, Malik R, Rasekh D, Ansari A, Corriveau RA, Ehrlich AR, Wang C, Ayers E. Non-literacy biased, culturally fair cognitive detection tool in primary care patients with cognitive concerns: a randomized controlled trial. Nat Med. 2024 Aug;30(8):2356-2361. doi: 10.1038/s41591-024-03012-8. Epub 2024 Jun 4. PMID 38834847
- [Derived] Chalmer R, Ayers E, Weiss EF, Malik R, Ehrlich A, Wang C, Zwerling J, Ansari A, Possin KL, Verghese J. The 5-Cog paradigm to improve detection of cognitive impairment and dementia: clinical trial protocol. Neurodegener Dis Manag. 2022 Aug;12(4):171-184. doi: 10.2217/nmt-2021-0043. Epub 2022 May 23. PMID 35603666
- See also: The Consortium for Detecting Cognitive Impairment, Including Dementia — https://www.detectcid.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5-Cog | Health Literacy & Grip Assessment
Started | 599 | 602
Completed | 592 | 600
Not Completed | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-Cog | Health Literacy & Grip Assessment | Total
Number analyzed (Participants) | 599 | 602 | 1201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 599 | 602 | 1201
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.88 (6.38) | 72.64 (6.67) | 72.76 (6.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 431 | 434 | 865
  Male | 168 | 168 | 336
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 323 | 344 | 667
  Not Hispanic or Latino | 275 | 258 | 533
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 13 | 10 | 23
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 305 | 280 | 585
  White | 59 | 59 | 118
  More than one race | 33 | 28 | 61
  Unknown or Not Reported | 183 | 220 | 403
Region of Enrollment [Number; unit: participants]
  United States | 599 | 602 | 1201
Education years [Mean (Standard Deviation); unit: years] | 11.24 (4.10) | 10.95 (4.26) | 11.09 (4.18)
Language of test administration [Count of Participants; unit: Participants]
  English | 339 | 342 | 681
  Spanish | 260 | 260 | 520

OUTCOME MEASURES:

1. Primary Outcome: New Occurrence in Dementia Care-A Composite Endpoint Including New Cognitive Diagnoses, Laboratory Investigations Related to Cognitive Impairment, New Dementia Prescriptions, and Cognitive Related Referrals.
Description: Dementia care is defined as the occurrence of any of the following endpoints following the screening visit. The endpoint is the number of participants who received 1 or more of the following orders:
  1. Any new diagnosis of dementia (relevant International Classification of Diseases (ICD)-10 codes) or Mild Cognitive Impairment (MCI) documented in the EMR.
  2. Tests ordered for reversible causes of cognitive impairment as recommended by the published guidelines of professional societies (i.e. thyroid function tests, B-12 level, Syphilis Panel, human immunodeficiency virus (HIV) test, computed tomography (CT) or Magnetic Resonance Imaging (MRI) scans) documented in the EMR.
  3. Any new prescriptions for dementia medications (i.e. Donepezil, Aricept, Memantine, Namenda, Rivastigmine, Exelon, Galantamine, Razadyne, Donepezil, or Namzaric) documented in the EMR.
  4. Referral for cognitive/dementia evaluation by specialists (i.e. Neurology, Geriatrics or Psychiatry) documented in the EMR.
Time Frame: 90 days after the participant is randomized
Measure: Count of Participants; unit: Participants
Arm/Group | 5-Cog | Health Literacy & Grip Assessment
Number analyzed (Participants) | 599 | 602
Participants | 111 | 41
Statistical Analysis 1: Comparison: 5-Cog vs Health Literacy & Grip Assessment; The estimate of odds ratio, its 95% confidence interval and p-value are obtained from logistic regression models which were used to examine the difference in dementia care outcomes between the intervention and control groups at 90 days post screening visit. Models are adjusted for age, sex, and years of education; Test type: Superiority; Odds Ratio (OR) = 3.43, 95% CI 2-sided [2.32 to 5.07]

2. Secondary Outcome: New Occurrence of in Health Care Utilization
Description: Utilization is defined in terms of emergency room visits and hospitalizations following the screening visit. The number of participants who went to the emergency room or had a hospitalization in the 6 months following the screening visit are presented in aggregate.
Time Frame: 6 months after the participant is randomized
Measure: Count of Participants; unit: Participants
Arm/Group | 5-Cog | Health Literacy & Grip Assessment
Number analyzed (Participants) | 599 | 602
Participants | 106 | 96
Statistical Analysis 1: Comparison: 5-Cog vs Health Literacy & Grip Assessment; The estimate of odds ratio, its 95% confidence interval and p-value are obtained from logistic regression models which were used to examine the difference in participants who were hospitalized or visited an ER 6 months post screening visit; Test type: Superiority; Odds Ratio (OR) = 1.133, 95% CI 2-sided [0.837 to 1.534]

3. Other Pre Specified Outcome: Cost-effectiveness
Description: Medicare payments for health care utilization will be valued. Costs will be divided into fixed and variable costs and by the screening and follow-up phases. Total costs will be estimated for health care utilization and reimbursement data captured by the EMR.
Time Frame: 6 months after the participant is randomized
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Health Care Utilization
Description: Utilization is defined in terms of specialty visits, emergency room visits, and hospitalizations following the screening visit.
Time Frame: 12 months after the participant is randomized
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Cost-effectiveness
Description: as for outcome 3
Time Frame: 12 months after the participant is randomized
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 90 days
Description: Participants were monitored specifically for study-related adverse events (i.e., medical symptoms, anxiety, depressive symptoms, etc.) that occurred in the 90 days following the assessments.
Arm/Group | 5-Cog | Health Literacy & Grip Assessment
All-Cause Mortality (participants affected / at risk) | 0/599 | 0/602
Serious Adverse Events (participants affected / at risk) | 0/599 | 0/602
Other Adverse Events (participants affected / at risk) | 0/599 | 0/602

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT03816644/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT03816644/ICF_001.pdf